CLINICAL TRIAL: NCT02793037
Title: A Proof of Concept for All-ceramic Zirconia Resin Bonded Bridges for Canine, Premolar and Short Span Posterior Teeth Official Title:
Brief Title: A Proof of Concept for All-ceramic Zirconia Resin Bonded Bridges for Canine, Premolar and Short Span Posterior Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr Michael G. Botelho, Clinical Associate Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW 15-205
Record Dates: First submitted 2016-05-20; First posted 2016-06-08 (Estimated); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Missing Teeth
Keywords: zirconia; resin bonded bridge
MeSH Terms: conditions — Anodontia

ARMS (1):
- A proof of concept of using zirconia bonded bridge (Experimental)
  Interventions: Device: Zirconia resin bonded bridge

INTERVENTIONS:
Device: Zirconia resin bonded bridge

SUMMARY:
Trial Design - Objectives and Purpose The aim of this study is to perform a proof of concept for the successful retention and outcome measures of zirconia RBBs for the replacement of missing canine or posterior teeth (6-8mm span) and that they will exhibit similar survival rates (95%) as metal ceramic RBBs over 3 years and short term (Botelho 2006).

The use of monolithic extra-coronal zirconia RBBs in the posterior region does not appear to have been reported in the literature (A search pf Pub Med and Google Scholar has not shown any similar studies that have been published - pubmed.gov; Keywords: "zirconia", "resin", "clinical" assessed on 17/10/2015 AND google scholar; Keywords: "zirconia", "resin bonded fixed partial denture", "resin bonded fixed dental prosthesis", "Maryland", "resin bonded bridge" "posterior", "clinical") In addition, currently there appear to be no clinical trials planned or finished in this area (clinicaltrial.gov; Keywords: "zirconia", "resin" assessed on 17/10/2015) using zirconia RBBs in the posterior region. This reveals that there is a gap in the literature on the use of zirconia for replacing posterior teeth with such prostheses.

The primary outcome measures would be: success ie. prosthesis retention ie. does not fall out

The secondary outcome measures would be:

* complications of the prosthesis such as tipping, drifting or fracture.
* patient centered outcomes (satisfaction and oral health related quality of life) on the RBBs The hypothesis is that 2-unit cantilevered zirconia RBBs will be as successful as current data on 2-unit cantilevered metal-ceramic RBBs from this centre and that there will be no difference in the patient centered outcomes.

The Primary review appointments will be at 1, 6, 12, 24 and 36 months. However, longer term follow up will be performed and this centre has experience of such long term studies (9.5 years - Botelho 2014).

A randomized clinical trial (RCT) comparing to metal-ceramic RBBs will NOT be performed as the 5-year success rate of both metal-ceramic (Botelho 2006) and anterior zirconia (Sasse 2014) prosthesis were higher than 95% and this small differences would mean an unattainable large sample size in an equivalence test (Burns 2001).

Significance and implications Zirconia has significant strength and greater stiffness than base metal alloys and displays clinical outcomes comparable to metal-ceramic conventional crowns and bridges (Heintze 2010, Sailer 2007). Well polished zirconia has been observed to have lower wear rates than porcelain (Stober 2014) Zirconia RBBs for posterior tooth replacement will offer an esthetic and biocompatible treatment option to patients over the traditional ceramic-metal RBBs. It is anticipated that patient demand for this would be high as these prostheses should be as successful (retentive).

These results would re-write established dental prosthodontics textbooks and this would be the first centre to report on the routine use of a 2-unit extracoronal all-zirconia RBB for the replacement of missing posterior teeth.

Research plan and methodology The sample pool would be obtained from patients presenting at the Prince Philip Dental Hospital, University of Hong Kong and who request and need replacement of one or more missing teeth.. They will be clinically assessed for eligibility and invited to participate with written consent in the study. After treatment they will be reviewed up to a 3rd year endpoint of the study. Further review beyond this will be undertaken.

ELIGIBILITY:
Inclusion Criteria:

* • The patient is over 18 years old.

  * A minimum of one single missing canine, premolar, or molar tooth raging in length from 6-8 mm as judged by the span between the contact points of the adjacent teeth from study models..
  * After discussion of treatment options, and that RBB is the most suitable treatment option for them, they will be invited to participate in the study.
  * The patient will be rendered dentally fit ie. controlled dental disease - no active caries or periodontal disease
  * Have a minimum of 12 occluding pairs of natural teeth
  * They will have been informed on the nature of the study and signed consent forms agreeing to undertake treatment in the study.
  * Patients will be available to be reviewed at 1, 6, 12, 24, and 36 months and longer.

Exclusion Criteria:

* • Patients with active tooth decay.

  * Patients with uncontrolled periodontal disease. An RBB abutment with a probing depth greater than 5mm and bleeding on probing.
  * Patients with teeth missing opposite to the planned RBB.
  * Abutment tooth mobility of 2 or greater (Millers classification).
  * Patients with debilitating illnesses or complicating medical conditions.
  * Non-vital or root treated abutment teeth.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Zirconia bridge clinical retention/survival rate, that is the presence of the zirconia bridge in patients' mouth in review appointment and will be calculated as a percentage of the total bridges placed as well as presented in Kaplan Meier survival curve. | 3 years

SECONDARY OUTCOMES:
Patient satisfaction in terms of oral health related quality of life (OHrQoL) using Oral Health Impact Profile (OHIP) 49-items questionnaire | 3 years
Patient satisfaction in terms of bridge satisfaction in visual analogue scale (VAS) | 3 years
Complications/adverse outcome associated with Zr bridge reported by patient and detected by clinical assessors | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Oral Rehabilitation, Faculty of Dentistry, The University of Hong Kong, Hong Kong, Guangdong, China

REFERENCES:
- [Derived] Lam WYH, Lim TW, Yu Yon MJ, Chau JMH, Lai GCH, Wang DCP, Botelho MG. Posterior two-unit cantilevered zirconia resin-bonded fixed partial dentures: A 3-year prospective single-arm clinical trial. J Dent. 2024 Aug;147:105140. doi: 10.1016/j.jdent.2024.105140. Epub 2024 Jun 18. PMID 38901823